CLINICAL TRIAL: NCT01952834
Title: Effect of Probiotic Supplementation on Endothelial Function in Men With Coronary Artery Disease
Brief Title: Effect of Probiotic Supplementation on Endothelial Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00019610; FP00004156 (Other: CTSI Advancing a Healthier Wisconsin)
Record Dates: First submitted 2013-09-24; First posted 2013-09-30 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; probiotic; endothelial function; brachial artery; ntric oxide
MeSH Terms: conditions — Coronary Artery Disease | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GoodBelly Probiotic and Vancomycin (Experimental): Good Belly Probiotic 2.7 oz Daily x 6 weeks Followed by a 4 week wash out period and then, Vancomycin, a non absorbed antibiotic administered (250 mg four times daily) orally for 10 days
  Interventions: Dietary Supplement: GoodBelly Probiotic; Drug: Vancomycin

INTERVENTIONS:
Dietary Supplement: GoodBelly Probiotic — GoodBelly Probiotic 2.7 oz Daily x 6 weeks. Followed by a 4 week wash out period and then, Vancomycin, a non absorbed antibiotic administered (250 mg four times daily) orally for 10 days
Drug: Vancomycin — GoodBelly Probiotic 2.7 oz Daily x 6 weeks. Followed by a 4 week wash out period and then, Vancomycin, a non absorbed antibiotic administered (250 mg four times daily) orally for 10 days

SUMMARY:
The study is being performed to determine whether probiotics (GoodBelly) improves blood vessel function.Probiotics similar to yogurt are living micro-organisms (beneficial to its host) the lives in the intestine. Patients who have coronary artery disease will be enrolled in this study. The research results will be used to determine if the type of bacteria present in the intestines play a role in the pathogenesis of cardiovascular disease. Patients with coronary artery disease will be enrolled for up to 12 weeks. Patients will take the probiotic for 6 weeks. Following the 6 week period there is a washout period of 4 weeks, and an optional antibiotic study called vancomycin. Patients will take the vancomycin for 10 days. Blood vessel function will be measured by ultrasound before and after the probiotic supplement and vancomycin antibiotic. Blood will also be taken before and after to evaluate for markers of inflammation.

DETAILED DESCRIPTION:
We plan to recruit 20 patients, men with coronary artery disease, for this single center, interventional trial with the Probiotic-GoodBelly followed by Vancomycin. The study includes 6 total visits. Subjects who pass a phone screen will be invited to a screening visit for study eligibility (Visit 1) Informed consent will be reviewed; a unique study number will be assigned once written informed consent is obtained (no subject will be assigned more than 1 allocation number); relevant participant medical history will be recorded including currently prescribed medications; anthropometric measurements will be taken (height, weight, and waist circumference in metric units) and blood pressure will be recorded (measured in triplicate and averaged). Subjects will be allowed to take their blood pressure medication on the morning of their screening visit, but not the mornings of any of the other study visits to limit the acute influence of these medications on endothelial function. If the potential participant qualifies for the study, he will return 1 week after the screen for a study visit(Visit 2) where he will turn in his stool sample, undergo initial tests of endothelial function and receive 3 week supply of GoodBelly Probiotic. After 3 weeks he will have to return (Visit 3) for another 3 week supply of his probiotic. After a total of 6 weeks of taking the probiotic he will have to return (Visit 4) with his stool sample. He will be asked to fast for 6-8 hours prior to the visit to limit the acute dietary influences on vascular endothelial function. During Visit 4, endothelial function will determined by brachial artery reactivity testing His stool samples will be collected and blood samples will also be taken at this visit for systemic measurements inflammatory markers. If he agrees to the optional Vancomycin study. He will return after 4 weeks for (Visit 5). He will be asked to fast for 6-8 hours prior to the visit to limit the acute dietary influences on vascular endothelial function. At Visit 5, endothelial function will determined by brachial artery reactivity testing His stool samples will be collected and blood samples will also be taken at this visit for systemic measurements inflammatory markers. He will then be given a 10 day supply of vancomycin. After 10 days he will return (Visit 6) with his stool sample. At Visit 6, endothelial function will determined by brachial artery reactivity testing . His stool samples will be collected and blood samples will also be taken at this visit for systemic measurements inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40-75 years old
2. Male sex
3. History of known coronary artery disease (by either history of myocardial infarction, angiogram demonstrative >=50% stenosis in at least 1 major epicardial coronary artery, or a previous stress test that showed evidence of ischemia that has not been revealed to be a false positive test by angiography)

Exclusion Criteria:

1. Unstable angina or myocardial infarction by history, ECG, and/or enzymatic criteria within 1 month of enrollment.
2. Left ventricular dysfunction as defined by an left ventricular ejection fraction documented as < 45% within 1 year of enrollment by an echocardiogram, MRI, or nuclear imaging.
3. Uncontrolled hypertension with a blood pressure greater than 170/100 mmHg at the screening visit.
4. Known history of chronic renal insufficiency, liver dysfunction, or cancer besides non-melanoma skin carcinomas or localized prostate cancer requiring systemic treatment within five years of enrollment.
5. Known history of cognitive impairment or inability to follow study procedures
6. Patient with an implanted defibrillator or permanent pacemaker on with the potential participant is known to rely upon for greater than 50% of ventricular depolarizations.
7. Patients who received probiotics, prebiotics, and antibiotics in the last 12 weeks.
8. Patients with dosing changes of vasoactive medications and 3-hydroxy-3-methylglutaryl-coenzyme A reductase inhibitors in the 6 weeks prior to enrollment.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Widlansky, MD, Principal Investigator — Medical College of Wisconsin; John Baker, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwauke, Wisconsin, United States

REFERENCES:
- [Derived] Malik M, Suboc TM, Tyagi S, Salzman N, Wang J, Ying R, Tanner MJ, Kakarla M, Baker JE, Widlansky ME. Lactobacillus plantarum 299v Supplementation Improves Vascular Endothelial Function and Reduces Inflammatory Biomarkers in Men With Stable Coronary Artery Disease. Circ Res. 2018 Oct 12;123(9):1091-1102. doi: 10.1161/CIRCRESAHA.118.313565. PMID 30355158

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GoodBelly Probiotic and Vancomycin
Started | 21
Completed | 20
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | GoodBelly Probiotic and Vancomycin
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
History of Hypertension [Number; unit: participants]
  Hypertensive | 11
  Non-Hypertensive | 10

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Flow Mediated Dilation
Description: A measurement of endothelial function in humans that reports the percent change in brachial artery diameter to a flow stimulus in the arm induced by 5 minutes of occlusion of flow to the arm. It is measured as the percent change from baseline diameter.
Time Frame: % Change before and after 6 weeks of daily Probiotic
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GoodBelly Probiotic and Vancomycin
Number analyzed (Participants) | 20
percent change | 1.2 (1.6)

2. Primary Outcome: Brachial Artery Flow Mediated Dilation
Description: Flow Mediated Dilation is measured as the percent change in brachial artery diameter as measured by high resolution ultrasound based on arterial diameter prior to and following 5 minute flow occlusion to the forearm . We measured the percent change in brachial diameter before vancomycin was started and again 10 days after vancomycin
Time Frame: Change before and after 10 days of Vancomycin, approximately 12 weeks from baseline
Population: Subgroup analyzed who volunteered to have vancomycin
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GoodBelly Probiotic and Vancomycin
Number analyzed (Participants) | 13
percent change | -0.2 (2.0)

3. Secondary Outcome: Interleukin 8
Description: Circulating cytokine measured in the plasma
Time Frame: Change before and after 6 weeks of daily Probiotic
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | GoodBelly Probiotic and Vancomycin
Number analyzed (Participants) | 18
pg/mL | -3.5 (1.3)

4. Secondary Outcome: Interleukin-12
Description: This is a circulating plasma cytokine
Time Frame: Change before and after 6 weeks of probiotic
Population: Subjects with plasma samples available pre and post probiotic supplementation
Measure: Mean (Standard Error); unit: pg/mL
Groups:
- Probiotic Supplementation: The measurement of IL-2 represents the change in IL-12 +/- standard deviation of the change following 6 weeks of probiotic supplementation.
Arm/Group | Probiotic Supplementation
Number analyzed (Participants) | 17
pg/mL | -10.4 (3.9)

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected over the 2 years of the open trial
Description: The categorization scheme A) Severity: 1) Mild 2) Moderate 3) Severe B) Expectedness 1) Expected- those consistent with the protocol in nature, severity, or frequency or 2) Unexpected C) Attribution 1) Unrelated to Protocol 2) Possibly Related to the Protocol 3) Probably Related to the Protocol 4) Definitely Related to the Protocol
Arm/Group | GoodBelly Probiotic and Vancomycin
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GoodBelly Probiotic and Vancomycin (N=21)
Stroke (Nervous system disorders) | 1 (1) — 1 participant suffered a stroke while on probiotic. In light of his known vascular disease a stroke is an event that could be reasonably expected. The event was judged as serious, not expected, and unrelated to the study protocol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No